CLINICAL TRIAL: NCT02667964
Title: FGF-21 During Physical Exercise in Patients With Type 1 Diabetes Mellitus, Type 2 Diabetes Mellitus and Healthy Controls
Brief Title: FGF-21 and Exercise in Relation to Insulin Secretion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Knut Mai, FGF-21 and Exercise, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FGF-Exercise
Record Dates: First submitted 2015-11-24; First posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy controls (Other): Spiroergometry
  Interventions: Other: spiroergometry
- Patients with T2DM (Other): Spiroergometry
  Interventions: Other: spiroergometry
- Patients with T1DM (Other): Spiroergometry
  Interventions: Other: spiroergometry

INTERVENTIONS:
Other: spiroergometry — Spiroergometry on a bicycle ergometer

SUMMARY:
FGF-21 and insulin are key hormones in the regulation of glucose metabolism. Furthermore, both hormones are influenced by physical activity. The following hypothesis will be tested: FGF-21 is regulated insulin-dependent during exercise.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a metabolic disorder characterized by rising global importance. In Germany alone, more than seven million people are being treated currently. T2DM is characterized by permanently elevated blood glucose levels, based on insulin resistance and followed by associated beta cell failure. In our previous work the investigators could already shown that increased FGF-21 levels are accompanied by an increased risk of T2DM. Physical activity is essential in the treatment and the prevention of T2DM. Interestingly, it was shown that acute physical exercise was leading to decreased insulin levels and increased FGF-21 values. In this study the effects of acute physical activity on FGF-21 values should be investigated in 3 groups: a) Healthy volunteers b) persons with T2DM c) persons with T1DM.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers,persons with T2DM, persons with T1DM

Exclusion Criteria:

* Patients with contraindications to an exercise ECG or spirometry be excluded from participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
FGF-21 change after physical activity | FGF-21 before and 1 h after spiroergometry

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bobbert, Dr, Principal Investigator — Charité
Locations (1):
- Charité, Berlin, State of Berlin, Germany